CLINICAL TRIAL: NCT03712657
Title: Multi-center Research Manual for the Perioperative Application of Enhanced Recovery After Surgery in Pediatric Acute Appendicitis
Brief Title: ERAS for Pediatric Acute Appendicitis
Acronym: EPAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Feng Jiexiong (Other)
Responsible Party: Sponsor-Investigator, Feng Jiexiong, professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJH
Record Dates: First submitted 2018-10-07; First posted 2018-10-19 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Pediatric Disorder; Complicated Appendicitis
Keywords: ERAS; Pediatric surgery; Emergency; Both of systolic and diastolic will be measured
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Experimental): interventions: 1.preoperative pain control; 2.avoiding application of ureter; 3.avoiding application of gastric tube; 4.avoiding application of irrigation; 5.avoiding application of drainage; 6.early exercising postoperatively; 7.early oral feeding postoperatively; 8.early discharging.
  Interventions: Combination Product: ERAS
- control group (No Intervention): normal treatment

INTERVENTIONS:
Combination Product: ERAS — 1. preoperative pain control;
  2. avoiding application of ureter;
  3. avoiding application of gastric tube;
  4. avoiding application of irrigation;
  5. avoiding application of drainage;
  6. early exercising postoperatively;
  7. early oral feeding postoperatively;
  8. early discharging.
  Arms: ERAS group

SUMMARY:
This multicenter, prospective randomized controlled study is designed to applicate perioperative Enhanced recovery after surgery (ERAS) management for children with acute complicated appendicitis, the aim is to promote postoperative recovery, shorten the hospital length of stay, and reduce the incidence of postoperative complications.

DETAILED DESCRIPTION:
The purpose of this study is through multi-center prospective RCT research, to discuss the application of ERAS in children with acute complicated appendicitis, including its preoperative rehydration, postoperative analgesia, preoperative and postoperative antibiotics application, as well as the discharge standards and so on. The major outcome is whether it can reduce the length of stay in hospital (LOS), secondary outcomes are included the incidence of postoperative complications and postoperative readmission rate, etc.

ELIGIBILITY:
Inclusion Criteria:

* ages<14; no gender limitation;
* Alvarado scores ≥7;
* preoperative radiography examination indicated complicated appendicitis;
* Patients or their legal representatives have signed "informed consent"

Exclusion Criteria:

* complicated life-threatening disease;
* perioperative exploration not appendicitis;
* Recently participated in other clinical trials within 3 months;
* Researchers found not fit to participate in this trial for any condition

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 893 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
length of stay | through study completion, an average of 7 days
  less hospital length of stay

SECONDARY OUTCOMES:
first time for postoperative feeding | up to 72 hours
  earlier postoperative feeding
first time for postoperative exercising | 1-2 days
  earlier postoperative exercising
rate of postoperative complication | 1 months
  less postoperative complication
rate of re-operation | 1 months
  less rate of re-operation
rate of re-admission | 1 months
  less rate of re-admission

CONTACTS AND LOCATIONS:
Overall Officials: Jiexiong Feng, MD, Principal Investigator — Tongji Hospital, HUST, China
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data for all primary and secondary outcome measures will be made available.